CLINICAL TRIAL: NCT04008017
Title: The Role of Eosinophilic Cationic Protein as a Biomarker in Diagnosis of Acute Exacerbation of Chronic Obstructive Pulmonary Disease at Assiut University Hospital
Brief Title: Eosinophilic Cationic Protein as a Biomarker in Diagnosis of Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: COPD-ECP
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stable Chronic obstructive pulmonary disease: clinical features of Chronic obstructive pulmonary disease and associated spirometry compatible with the GOLD criteria (Forced expiratory volume 1/ Forced vital capacity <70%) post bronchodilator
  Interventions: Diagnostic Test: Eosinophilic Cationic Protein biomarker
- acute exacerbation of Chronic obstructive pulmonary disease: patients developed fever, increased dyspnea and sputum production plus the clinical features of Chronic obstructive pulmonary disease and associated spirometry compatible with the GOLD criteria (Forced expiratory volume 1/ Forced vital capacity <70%) post bronchodilator
  Interventions: Diagnostic Test: Eosinophilic Cationic Protein biomarker

INTERVENTIONS:
Diagnostic Test: Eosinophilic Cationic Protein biomarker — 3 ml blood for serum sample for estimation of Eosinophilic Cationic Protein biomarker level using ELISA

SUMMARY:
Chronic obstructive pulmonary disease is a type of obstructive lung disease characterized by long-term breathing problems and poor airflow. It is changed to acute exacerbation of Chronic obstructive pulmonary disease when respiratory symptoms worsen, beyond normal day-to-day variations, severely enough that changes in medication are required.

Inflammation is a core feature of acute exacerbation of Chronic obstructive pulmonary disease since it gives insight into the pathological changes causing an exacerbation. Eosinophils may play a significant role in airway inflammation in some patients with Chronic obstructive pulmonary disease.

Previous studies have indicated that eosinophilic airway inflammation is also associated with the development of severe acute exacerbation of Chronic obstructive pulmonary disease. Eosinophilic Cationic Protein has various biological activities, including antibacterial, antiviral, antiparasitic and neurotoxic functions, and it contributes to the regulation of fibroblast activity. Eosinophilic Cationic Protein also induces airway mucus secretion and interacts with the coagulation and complement systems. Eosinophilic Cationic Protein has been developed as a marker for eosinophilic disease and quantified in biological fluids including serum, bronchoalveolar lavage and nasal secretions. It is found in diseases such as allergic asthma and allergic rhinitis but also occasionally in other diseases. Only activated eosinophil granulocytes release the granule content and therefore the determination of Eosinophilic Cationic Protein concentration is a considerably more specific indicator of eosinophil inflammation than eosinophil granulocyte count in peripheral blood as serum Eosinophilic Cationic Protein levels increase during acute exacerbation of Chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* clinical features of Chronic obstructive pulmonary disease
* spirometry compatible with the GOLD criteria (Forced expiratory volume 1/ Forced vital capacity <70%) post bronchodilator.

Exclusion Criteria:

* Patients with bronchial asthma
* Asthma -Chronic obstructive pulmonary disease overlap syndrome
* Atopic patients
* Pneumothorax
* Congestive heart failure
* Cancer of any kind
* A history of major surgery in the preceding 4 weeks.
* Patients undergoing mechanical ventilation or presenting with azotaemia (serum creatinine >1.5 mg/dl).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed diagnosis of Chronic obstructive pulmonary disease and acute exacerbation of Chronic obstructive pulmonary disease based on Gold guidelines, at the Chest Department and Respiratory Intensive Care Unit and chest outpatient clinic at Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The mean difference in the level of Eosinophilic Cationic Protein biomarker in the two study groups | 3 months
  measurement by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt